CLINICAL TRIAL: NCT01252030
Title: Impact of Telemonitoring Intervention on Physical Activity, CVD Risk Factors, During Phase 2-3 Cardiac Rehabilitation
Brief Title: Telemonitoring During Phase 2-3 Cardiac Rehabilitation
Acronym: TeleRehabII
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Paul Dendale, dr, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Telemonitoring 2
Record Dates: First submitted 2010-12-01; First posted 2010-12-02 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Ischemic Heart Disease
Keywords: CAD, physical activity, rehabilitation, prevention
MeSH Terms: conditions — Myocardial Ischemia; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- intervention (Experimental): stimulation of physical activity by messages sent through e mail or SMS; in combination with monitoring of physical activity with physical activity monitors
  Interventions: Device: physical activity monitors
- control (Placebo Comparator): no stimulation of physical activity
  Interventions: Other: No physical activity monitors

INTERVENTIONS:
Device: physical activity monitors — physical activity monitors
  Arms: intervention
Other: No physical activity monitors — No physical activity monitors
  Arms: control

SUMMARY:
In this study, 80 coronary artery disease patients with successful coronary revascularisation (by CABG or PCI) will be included. Patients are excluded in case of: congestive heart failure, ICD or pacemaker, any disability limiting exercise participation.

These patients are attending phase 2-3 cardiac rehabilitation, and have completed 6 weeks of rehabilitation. Next, subjects are randomly assigned to a control group or an intervention group.

Outcome parameters: physical activity, exercise capacity, blood glucose, insulin level and lipid profile, body weight and waist circumference, cardiovascular morbidity and mortality.

Hypothesis: telemonitoring of physical activity will increase physical activity, and improve cardiovascular disease risk factors, in CAD patients attending phase 2-3 cardiac rehabilitation.

DETAILED DESCRIPTION:
We included patients that suffered from an acute coronary syndrome for which a percutaneous coronary intervention or coronary artery bypass graft was performed.

All patients had access to a computer with internet connection.

Patients that (i) were more than 80 years old, (ii) had an implantable cardioverter defibrillator or pacemaker, (iii) suffered from severe arrhythmias, or (iv) had persistent exertional ischaemia after revascularization therapy, were not invited to participate in this study. Patients with severe heart failure (NYHA class III and IV), or neurological or orthopaedic disability limiting their capability to exercise, were also excluded.

The study was a prospective randomized controlled trial, including an 18-week intervention. All patients were included after week six of their conventional phase II cardiac rehabilitation (CR). During phase II of conventional CR, all patients (those in the intervention and control group) were educated about the core components of CR including healthy nutrition, risk factor management (lipids, hypertension, weight, diabetes, and smoking), psychosocial management and physical activity counseling.

During the first six weeks of the intervention, patients in the intervention group continued exercising in the hospital's rehabilitation centre using an outpatient service, in combination with an exercise training program with telemonitoring support. Patients in the control group continued exercising in the hospital's rehabilitation centre using an out-patient service, without participating in the exercise training program with telemonitoring support. Starting from the seventh week in the study period, patients in the intervention group finished their phase II CR in the hospital's rehabilitation centre but continued their exercise training program with telemonitoring support; patients in the control group finished their phase II CR in the hospital's rehabilitation centre.

All patients underwent a maximal cardiopulmonary exercise test (CPET) and a clinical examination (with determination of waist circumference, blood pressure, body mass index) after randomization, and also during the sixth and 18th week of the Telerehab II study period. A fasting blood sampling was taken from all patients during the first and 18th week of the Telerehab II study period.

The hypothesis was that telemonitoring of physical activity will increase physical activity, and improve cardiovascular disease risk factors, in CAD patients attending phase 2-3 cardiac rehabilitation.

ELIGIBILITY:
Inclusion Criteria: CAD patients following phase 2-3 rehabilitation -

Exclusion Criteria: CHF, pacemaker, ICD, any disability limiting exercise participation

-

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Physical activity | every week

SECONDARY OUTCOMES:
exercise capacity | every 6 weeks
blood lipid profile, glucose and insulin level | every 6 weeks
mortality and morbidity | continuously

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Dendale, MD, PhD, Principal Investigator — University of Hasselt, Hasselt, Belgium
Locations (1):
- Jessa Hospital, Hasselt, Belgium